CLINICAL TRIAL: NCT07314723
Title: A Single Arm, Open-label, Multicenter, Phase II Clinical Study to Evaluate the Safety and Efficacy of 9MW2821 Combined With Toripalimab in Perioperative Patients With Urothelial Cancer
Brief Title: 9MW2821 Combined With Toripalimab in Perioperative Patients With Urothelial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-CP202
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: MIBC (Experimental)
  Interventions: Drug: 9MW2821; Drug: Toripalimab Injection
- Arm 2: High-risk UTUC (Experimental)
  Interventions: Drug: 9MW2821; Drug: Toripalimab Injection
- Arm 3: MIBC (Experimental)
  Interventions: Drug: 9MW2821; Drug: Toripalimab Injection

INTERVENTIONS:
Drug: 9MW2821 — 9MW2821, 1.25mg/kg, intravenous (IV) infusion
Drug: Toripalimab Injection — Toripalimab, 240mg, intravenous (IV) infusion

SUMMARY:
This is a single arm, open-label, multicenter phase II clinical study to evaluate the safety and efficacy of 9MW2821 combined with Toripalimab in perioperative patients with urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form approved by IEC.
* Male or female subjects aged ≥18 years old.
* ECOG status: 0 or 1.
* Histologically confirmed urothelial cancer.
* Imaging confirmed non-metastatic urothelial cancer (M0). Arm 1: MIBC, T2-4aN0-1. Arm 2: High-risk UTUC, N0. Arm 3: MIBC, T2-4aN0.
* Adequate tumor tissues submitted for test.
* Life expectancy for more than 12 weeks.
* Adequate organ functions.
* Proper contraception methods.
* Willingness to follow the study procedures.

Exclusion Criteria:

* Prior systemic anti-tumor therapy for urothelial cancer.
* Previously treated with PD-1/PD-L1 inhibitors or antibody-drug conjugates (ADCs).
* History of another malignancy within 3 years.
* History of autoimmune disease requiring systemic treatment within 2 years.
* History of clinically significant cardiac/cerebrovascular diseases or thrombosis within 1 year.
* Major surgery treated within 28 days; Cystoscopy/ureteroscopy biopsy or intravesical instillation therapy within 7 days.
* Peripheral neuropathy Grade ≥ 2.
* Any situations adding the risk of severe dry eye, active keratitis or corneal ulcer, etc.
* Active HBV/HCV/HIV infection, etc.
* Any other serious chronic or uncontrolled disease.
* Any live vaccines got within 28 days.
* Organ transplantation or allogeneic hematopoietic stem cell transplantation in the past.
* Any potent CYP3A4 inducers/inhibitors taken within 14 days.
* Known allergic sensitivity to any of the ingredients of the study drug.
* History of drug abuse or mental illness.
* Other conditions unsuitable into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR (Arm 1 and 2) | Up to 24 months
  Pathological complete response
cCR (Arm 3) | Up to 24 months
  Clinical complete response

SECONDARY OUTCOMES:
cORR | Up to 24 months
  Clinical objective response rate
Pathological downstaging rate (Arm 1 and 2) | Up to 24 months
DFS (Arm 1 and 2) | Up to 24 months
  Disease-free survival
Duration of clinical complete response (Arm 3) | Up to 24 months
PFS (Arm 3) | Up to 24 months
  Progression-free survival
OS | Up to 24 months
  Overall Survival
AE/SAE | Up to 24 months
  Adverse event, serious adverse event
Immunogenicity | Up to 24 months
  Anti-Drug Antibody (ADA) of 9MW2821
Nectin-4 and PD-L1 expression | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China